CLINICAL TRIAL: NCT01008085
Title: Randomized Comparison Between the STENTYS Self-expanding Coronary Stent and a Balloon-expandable Stent in Acute Myocardial Infarction - APPOSITION II
Brief Title: STENTYS Self-expanding Versus Balloon-expandable Stent in Acute Myocardial Infarction (AMI)
Acronym: APPOSITION ll
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stentys (Industry)
Responsible Party: Rene Spaargaren, Chief Medical Officer, STENTYS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST2009-02
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: STEMI
Keywords: STEMI; self-expandable; balloon-expandable
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-expanding stent (Experimental): Stentys stent
  Interventions: Device: Stentys coronary stent
- Balloon-expandable stent (Active Comparator): VISION/Driver
  Interventions: Device: Balloon-expandable stent

INTERVENTIONS:
Device: Stentys coronary stent — Self-expanding Nitinol stent
  Other Names: Self-expanding stent
  Arms: Self-expanding stent
Device: Balloon-expandable stent — VISION/Driver
  Other Names: VISION/Driver
  Arms: Balloon-expandable stent

SUMMARY:
Study hypothesis: the Stentys self-expandable Stent results into a better alignment of the struts to the vessel wall than a balloon-expandable stent within a few days after the procedure in acute myocardial infarction patients.

DETAILED DESCRIPTION:
Stent strut malapposition and stent underexpansion are a common phenomenon in AMI as a result of the changing anatomy after an AMI has occurred (thrombus dissolution, resolution of spasm) with the traditional balloon-expandable stent treatment. A self-expanding stent might lead to better stent strut apposition as it follows the contours of the vessel wall due to its self-expanding properties. This might result into better long term clinical outcomes like lower thrombosis rates.

ELIGIBILITY:
Inclusion Criteria:

1. Subject 18 years old.
2. Acute Myocardial Infarction defined as presence of at least two of the three items below:

   1. Detection of rise of cardiac biomarkers with a least one value above the 99th percentile of the upper reference limit (URL)
   2. Symptoms of ischaemia (chest pain) >20 minutes
   3. ECG changes indicative of new ischaemia: new ST-T changes (ST deviation ≥0.2mV precordial leads and/or ≥0.1mV limb leads) or new LBBB)
3. Reperfusion expected to be achieved within 12 hours from the onset of symptoms
4. Subject understands the nature of the procedure and provides written informed consent prior to the catheterization procedure.
5. Subject is willing to comply with specified follow-up evaluation and can be contacted by telephone.
6. Acceptable candidate for coronary artery bypass graft (CABG) surgery.
7. Male or non-pregnant female subject.

Angiographic Inclusion Criteria:

1. Reference vessel diameter >2.5mm and <4.0mm by visual estimate.
2. Target lesion <30mm in length by visual estimate

Exclusion Criteria:

1. Currently enrolled in another investigational device or drug study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
2. Coronary or cardiac intervention or major surgery of any kind within 30 days prior to the procedure.
3. Target vessel supplied by by-pass vessel
4. Patients on anticoagulation therapy (Coumadin)
5. Patient received thrombolytic therapy.
6. Myocardial infarction due to stent thrombosis, or infarct lesion at the side of a previously implanted stent
7. Cardiogenic shock
8. Any previous stent placement within 10mm (proximal or distal) of the target lesion.
9. Co-morbid condition(s) that could limit the subject's ability to participate in the study or to comply with follow-up requirements, or impact the scientific integrity of the study.
10. Concurrent medical condition with a life expectancy of less than 6 months.
11. Left ventricular ejection fraction (LVEF) <30% at the most recent evaluation.
12. Cerebrovascular accident or transient ischemic attack in the last 6 months.
13. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, or sensitivity to contrast media, which cannot be adequately pre-medicated.
14. Known serum creatinine level >2.5mg/dl or presence or history of renal failure

Angiographic Exclusion Criteria:

1. Unprotected left main coronary artery disease (obstruction greater than 50% in the left main coronary artery that is not protected by at least one non-obstructed bypass graft to the left anterior descending (LAD) or left circumflex (LCX) artery or a branch thereof).
2. Target vessel is excessively tortuous (two bends >90˚ to reach the target lesion).
3. Lesion location that is aorto-ostial or within 5mm of the origin of the LAD or LCX.
4. Target lesion is severely calcified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Stent strut apposition measured by optical coherence tomography (OCT) | 3 days after procedure

SECONDARY OUTCOMES:
Stent thrombosis | 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, Ph.D, Principal Investigator — ZNA, Middelheim, Belgium
Locations (1):
- C. Spaulding, Paris, France

REFERENCES:
- [Derived] Nakatani S, Onuma Y, Ishibashi Y, Karanasos A, Regar E, Garcia-Garcia HM, Tamburino C, Fajadet J, Vrolix M, Witzenbichler B, Eeckhout E, Spaulding C, Reczuch K, La Manna A, Spaargaren R, Capodanno D, Van Langenhove G, Verheye S, Serruys PW, van Geuns RJ. Incidence and potential mechanism of resolved, persistent and newly acquired malapposition three days after implantation of self-expanding or balloon-expandable stents in a STEMI population: insights from optical coherence tomography in the APPOSITION II study. EuroIntervention. 2015 Dec;11(8):885-94. doi: 10.4244/EIJY15M11_01. PMID 26549374
- [Derived] van Geuns RJ, Tamburino C, Fajadet J, Vrolix M, Witzenbichler B, Eeckhout E, Spaulding C, Reczuch K, La Manna A, Spaargaren R, Garcia-Garcia HM, Regar E, Capodanno D, Van Langenhove G, Verheye S. Self-expanding versus balloon-expandable stents in acute myocardial infarction: results from the APPOSITION II study: self-expanding stents in ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2012 Dec;5(12):1209-19. doi: 10.1016/j.jcin.2012.08.016. PMID 23257368